CLINICAL TRIAL: NCT01502176
Title: A Retrospective Register Study to Map the Frequency of Short Duration Atrial Fibrillation (AF) Among All Patients Admitted to Roskilde Sygehus in Denmark in 2010
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ole Dyg Pedersen, Medical doctor, Zealand University Hospital
Other Study IDs: MISP Proposal # 38233
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Type of Atrial Fibrillation; Medical History; Current Treatment; Complications
Keywords: atrial fibrillation; registry
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atrial fibrillation patients: All patients discharged from hospital with a diagnose of atrial fibrillation

SUMMARY:
Retrospective observational study of patients with atrial fibrillation admitted to Roskilde University Hospital in 2010.

DETAILED DESCRIPTION:
The study is a retrospective register study of all patients discharged from Roskilde Hospital with a primary diagnosis of AF in 2010. All data will be collected from the patient's medical records and only data from this specific admission will be recorded. No follow-up of the patients after discharge will be performed in this study. The study does not involve any randomization or any drug testing.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted and discharged with a diagnose of atrial fibrillation in 2010 at Roskilde University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Roskilde University Hospital, Roskilde, Copenhagen, Denmark